CLINICAL TRIAL: NCT02902692
Title: Examining the Effects of a Brief Mindfulness Based Intervention (BMBI) on Mood and Cognitive Functioning in an Older Adult Population
Brief Title: Mindfulness for Older Adults With Cognitive Concerns
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16/LO/0223
Record Dates: First submitted 2016-08-31; First posted 2016-09-16 (Estimated); Last update posted 2016-09-16 (Estimated); Status verified 2016-04

CONDITIONS: Mild Cognitive Impairment
Keywords: brief; mindfulness
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brief Mindfulness (Experimental): 45 minute brief mindfulness intervention (lead by study investigator) on day 1 followed by 7 days of 30 minute mindfulness practice at home (without study investigator)
  Interventions: Other: Brief Mindfulness

INTERVENTIONS:
Other: Brief Mindfulness — 15 minutes psycho-education about mindfulness and a small experiential exercise using a raisin. Following this, participants listen to a 30minute pre-recorded sitting meditation which encourages them to focus on their breath and the sounds around them. Participants will be randomly assigned to either receive the brief mindfulness intervention immediately or will be asked to wait one week before receiving the intervention.

SUMMARY:
The current study will examine the effects of a brief mindfulness based intervention (BMBI) on mood, memory and attention in comparison to a wait-list control (WLC) group. Participants for the study will be 90 adults aged 50 years and above who have presented at a memory clinic within SLaM NHS Trust with subjective cognitive concerns and/or those who have received a diagnosis of mild cognitive impairment (MCI) from their memory clinic.

DETAILED DESCRIPTION:
Participants will be randomly assigned to either the BMBI group or the WLC group. Those assigned to the BMBI group will complete a number of cognitive assessments and questionnaires at Time 1. They will then receive a 45 minute mindfulness intervention. Following this, they will be asked to practice mindfulness for 30 minutes per day for 7 days a week in their own homes. After 7 days, participants in the BMBI group will be invited to complete a paired set of cognitive assessments and questionnaires (Time 2). Participants in the WLC group will complete the same number of cognitive assessments and questionnaires as the BMBI group at Time 1. However, they will not receive the 45 minute mindfulness intervention nor will they be asked to practice it at home for 7 days. After 7 days, participants in the WLC group will be invited to complete a paired set of cognitive assessments and questionnaires (Time 2). After completion of the measures at Time 2, the WLC participants will then receive the 45 minute mindfulness intervention. All assessments, questionnaires and the intervention will be carried out either in a SLaM memory clinic or at participants own homes depending on level of mobility.

ELIGIBILITY:
Inclusion Criteria:People aged 50 years and older with subjective memory concerns (SMC) and/or those who meet criteria for amnestic mild cognitive impairment (MCI) who have been seen by one of the three SLAM memory services (i.e. Croydon Memory Service; Southwark and Lambeth Memory Service; and Lewisham Memory Service) in the past three months. Participants must be able to give informed consent to participate.

-

Exclusion Criteria: Diagnosis of dementia or multi-domain mild cognitive impairment, intellectual disability, current substance misuse, a current diagnosis of epilepsy or another neurodegenerative disorder (such as Parkinson's), a history of brain injury or stroke, a severe and enduring mental health disorder (e.g. severe depression or anxiety, personality disorder, schizophrenia, schizoaffective disorder, bipolar affective disorder), active suicidal ideation, severe sensory impairment that would significantly impair a person's ability to engage in the intervention.

-

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Test of Everyday Attention | Change in attention from Baseline to 1 Week
  The Test of Everyday Attention (TEA): Two subtests from the TEA (Robertson et al., 1994) will be used in the current study. Specifically, the Elevator Test will be used to measure sustained attention and the Visual Elevator Test will be used as a measure of attentional switching, and hence of cognitive flexibility. The TEA subtests are based on everyday life scenarios offering greater ecological validity. It has parallel forms which allow for repeat administration within short time periods reducing the impact of practice effects.

SECONDARY OUTCOMES:
Hospital Anxiety Depression Scale (HADS) | Change in anxiety and depression from Baseline to 1 Week
  The HADS consists of two subscales measuring depression and anxiety respectively. Each subscale consists of seven items and responses on the items are based on the relative frequency of symptoms over the past week using a four point Likert scale ranging from 0 (not at all) to 3 (very often indeed). Higher scores indicate higher levels of depression and anxiety, and scores of about 10 on each subscale indicate clinical significance.
Penn State Worry Questionnaire | Change in worry from Baseline to 1 Week
  Penn State Worry Questionnaire: The PSWQ is a 16-item measure of worry that has shown adequate internal consistency and convergent validity in elderly patients with GAD and controls( Beck et al., 1995 and Stanley et al., 2001). It uses a Likert rating from 1 (not at all typical of me) to 5 (very typical of me).
Short Form Health Survey | Change in quality of life from Baseline to 1 Week
  Short-Form Health Survey (SF-36): The physical and mental summary scores of the Short Form Health Survey (SF-36) (Van de Zee et al., 1993) are used to measure quality of life related to physical and mental aspects. The SF-36 is composed of 36 items measuring health across eight dimensions: physical functioning, social functioning, role limitations due to physical problems, role limitations due to emotional problems, pain, mental health, vitality, and general health perception. These eight subscales can be summarized into one physical and one mental component summary score. Each dimension score ranges from 0-100. Higher scores indicate better health-related quality of life.
The Trail Making Test Parts A&B | Change in executive functioning from Baseline to 1 Week
  The Trail Making Test (TMT; Army Individual Test Battery, 1944) is a commonly used neuropsychological test of visual attention and task switching. It consists of 2 parts: part A asks participants to connect a series of numbers in ascending order on a page, while part B requires participants to draw a line alternating between ascending numbers and letters. Part A is used primarily to capture processing speed whereas Part B requires more complex attention shifting, planning, and concentration, and is, thus, considered a valid index of executive control. The time taken to complete the task is the primary performance outcome
Digit Span Task | Change in working memory from Baseline to 1 Week
  Digit Span is a core working memory sub-test of the WAIS-IV (Wechsler, 2008). It requires participants to repeat a series of digits forwards and backwards with series ranging in length from 2 to 9 digits. This test also measures auditory sequential processing as the individual must recall auditory information and repeat it back aloud. The Digit Span subtest has revealed an average test-retest reliability of .82 (Wechsler, 2008b).
Letter-Number Sequencing Task | Change in working memory from Baseline to 1 Week
  Letter Number Sequencing is a subtest of the WAIS-IV (Wechsler, 2008) and is a measure of attention and short-term memory. Lemay et al. (2004) report test-retest reliability data of between .73 and .75 in a two-week interval in middle aged to elderly subjects suggesting it can be reliably used in repeated neuropsychological assessments.
The Cognitive Failures Questionnaire | Change in subjective cognitive concerns from Baseline to 1 Week
  The Cognitive Failures Questionnaire (Broadbent et al., 1982) will be used as a measure of subjective cognitive complaints. The CFQ has been shown to have acceptable internal consistency and retest reliability, and good face validity in a sample of older adults (Knight et al., 2004).
The Five Facet Mindfulness Questionnaire (FFMQ) | Change in mindfulness from Baseline to 1 Week
  The Five Facet Mindfulness Questionnaire (FFMQ): The FFMQ (Baer et al., 2006) assesses five components of mindfulness: observing, describing, acting with awareness, non-judging of inner experience, and non-reactivity to inner experience. It has been shown to have good internal consistency (Baer et al., 2006) and adequate construct validity (Baer et al., 2008).
Ruminative Response Scale of the Response Styles Questionnaire | Change in rumination from Baseline to 1 Week
  Ruminative Response Scale of the Response Styles Questionnaire (RRS of RSQ; Nolen-Hoeksema & Morrow, 1991). The RRS will be administered to assess participants' tendencies to ruminate in response to their symptoms of negative emotion. The RRS includes 22 items in response to depressed mood that are self-focused (e.g., "I think why do I always react this way?"), symptom focused (e.g., "I think about how hard it is to concentrate"), and focused on the possible consequences and causes of mood (e.g., "I think I won't be able to do my job if I don't snap out of this"), which participants rate on a scale from 1 (never) to 4 (always). Total scores range from 22 to 88 with higher scores indicating greater rumination.
Self-Compassion Scale Short-Form | Change in self-compassion from Baseline to 1 Week
  Self-Compassion Scale Short-Form (SCS-SF): The SCS-SF (Raes, Pommier, Neff, & Van Gucht, 2011) measures self-compassion and it has the following sub-scales: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification. Participants have to rate how often they behave in a stated manner (e.g., "When I'm going through a very hard time, I give myself the caring and tenderness I need") in a scale from 1 (almost never) to 5 (almost always). Total scores range from 12 to 60 with higher scores indicating greater self-compassion
CORE-10 | Change in general psychological functioning from Baseline to 1 Week
  CORE-10. The CORE-10 is a short, 10 item version of the CORE-OM, a standard measure of psychological distress
Discharge Satisfaction Questionnaire | Post-treatment
  The Discharge Satisfaction Questionnaire, (a standard service measure used within the MHOA CAG) will be completed by both the mindfulness and WLC group at post-intervention only to evaluate service satisfaction and the acceptability of the mindfulness intervention

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Gould, PhD,DClinPsy, Principal Investigator — King's College London
Locations (1):
- South London and Maudsely NHS Memory Services, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No